CLINICAL TRIAL: NCT05805787
Title: The Effect of Acupressure on Constipation Symptoms in Elderly
Brief Title: Acupressure for Constipation in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Yalova (Other)
Collaborators: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Yalova Uni.
Record Dates: First submitted 2023-03-26; First posted 2023-04-10 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Constipation
Keywords: elderly; defecation; laxatives; old age homes
MeSH Terms: conditions — Constipation | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: randomized, pretest-posttest control group study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): Acupressure will be applied to the elderly in the experimental group once a day, 5 days a week (Monday-Friday) for a week. The application will last for 2 weeks. A total of 10 sessions of acupressure will be applied. Acupressure application will be applied by researchers who have been trained and certified on this subject. While the elderly are in supine position, pressure will be applied to each acupressure point, respectively, Tianshu (ST25), Guanyuan (CV4) and Hegu (LI4) for 2 minutes for a total of 6 minutes.
  Interventions: Other: Acupressure
- Control group (No Intervention): No intervention will be applied

INTERVENTIONS:
Other: Acupressure — Acupressure will be applied to the elderly in the experimental group once a day, 5 days a week (Monday-Friday) for a week. The application will last for 2 weeks. A total of 10 sessions of acupressure will be applied. Acupressure application will be applied by researchers who have been trained and certified on this subject. While the elderly are in supine position, pressure will be applied to each acupressure point, respectively, Tianshu (ST25), Guanyuan (CV4) and Hegu (LI4) for 2 minutes for a total of 6 minutes.
  Arms: Acupressure group

SUMMARY:
This study will carried out to determine the effect of acupressure applied to Tianshu (ST25), Guanyuan (CV4) and Hegu (LI4) acupuncture points for a total of 6 minutes, two to each point, on the symptoms of constipation in the elderly people receiving institutional care.

DETAILED DESCRIPTION:
In a randomized controlled study will be evaluated the effect of acupressure application on constipation symptoms in the elderly people receiving institutional care. The study population will be conducted of 193 elderly individuals living in a Nursing and Rehabilitation Center under the Directorate of Family, Labor and Social Services in a province of Turkey. After explaining the purpose of the study and obtaining written consent from the patients, those with constipation will be determined. Those with constipation will be determined by applying The Patient Identification Form, Mini-Cog© Test, Constipation Diagnosis Form to the entire population. The sample of the study will consist of all patients who meet the inclusion criteria and who are willing to participate in the study. The sample size calculated using a t-test in independent samples with the G Power 3.1.3 software. In a randomized controlled study by Abbasi et al. (2019), it was seen that the effect size of acupressure on constipation was 0.99. When a single direction calculation was performed with a 95% confidence interval, 80% power, a ratio of 1:1 for Intervention and Control group, and a strong effect size (0.80), it was determined that it was necessary to choose a minimum of 21 patients for each group, that is, a total of 42 patients. Considering that there may be losses in the application and follow-up period, the number of samples will be increased by 10% and 23 people will be included in each group. The patients enrolled in the study will be divided into intervention and control groups using the previously prepared randomization checklist. After the Intervention and Control group is determined, all patients will be followed for a total 10 days and the Bristol Stool Scale and Constipation Assessment Scale will be applied daily. Acupressure will be applied to the elderly in the experimental group once a day, 5 days a week (Monday-Friday) for a week. The application will last for 2 weeks. A total of 10 sessions of acupressure will be applied. Acupressure application will be applied by researchers who have been trained and certified on this subject. While the elderly are in supine position, pressure will be applied to each acupressure point, respectively, Tianshu (ST25), Guanyuan (CV4) and Hegu (LI4) for 2 minutes for a total of 6 minutes. No attempt will be made to the control group. All patients will be followed during the application (14 days) and for 10 days after the application and the Bristol Stool Scale and Constipation Assessment Scale will be applied daily. After the data is coded and transferred to the computer environment, it will be evaluated with the SPSS 21.0 program. Pre-test post-test results of the Intervention and Control groups will be analyzed for variance in the t-test and repeated measurements applied in independent groups. Confidence interval for statistical significance will be set as <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 and over,
* Experiencing two or more of the Rome IV criteria
* Not following a special nutrition program
* Not using laxatives

Exclusion Criteria:

* Have a communication problem
* Having high cognitive impairment (according to the Mini-Cog test)
* Addicted to bed
* Having musculoskeletal problems (eg amputation of the acupuncture site)
* Having received acupressure / acupuncture treatment up to 8 weeks before the study
* Having skin problems at acupressure points (eg, skin rash, infection)
* History of gastrointestinal disorders such as irritable bowel syndrome, rectal prolapse, anal fissure, volvulus, and bowel obstruction

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Constipation Assessment Scale | Change from Baseline symptoms of constipation at 24 days
  It will be used to evaluate the symptoms of constipation.Constipation Assessment Scale prepared according to the Rome IV criteria for the diagnosis of constipation. According to the criteria, 2 or more of the following symptoms must have started at least 6 months ago and continued for the last 3 months.
  i. Straining more than 25% of defecations. ii. Lumpy or hard stools (The Bristol Stool Form Scale type 1 or 2) more than 25% of defecations.
  iii. Sensation of incomplete evacuation more than one-fourth (25%) of defecations.
  iv. Sensation of anorectal obstruction/blockage more than one-fourth (25%) of defecations.
  v. Manual maneuvers to facilitate more than one-fourth (25%) of defecations. vi. Fewer than three spontaneous bowel movements per week
Bristol Stool Scale | Change from Baseline symptoms of constipation at 24 days
  It will be used to determine the characteristics of the stool. This helps assess how long the stool has spent in the bowel. Types 1 and 2 indicate an unusually hard stool and constipation. types 6 and 7 are unusually loose and may indicate diarrhea. A normal stool should be a type 3, 4, and 5.

SECONDARY OUTCOMES:
Number of Defecation | Change from baseline number of defecations at 24 days
  24-day total number of defecations

CONTACTS AND LOCATIONS:
Overall Officials: Esra Usta, PhD, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbasi P, Mojalli M, Kianmehr M, Zamani S. Effect of acupressure on constipation in patients undergoing hemodialysis: A randomized double-blind controlled clinical trial. Avicenna J Phytomed. 2019 Jan-Feb;9(1):84-91. PMID 30788281
- [Result] Ho MH, Chang HCR, Liu MF, Yuan L, Montayre J. Effectiveness of acupoint pressure on older people with constipation in nursing homes: a double-blind quasi-experimental study. Contemp Nurse. 2020 Oct-Dec;56(5-6):417-427. doi: 10.1080/10376178.2020.1813042. Epub 2020 Sep 18. PMID 32814493